CLINICAL TRIAL: NCT05725330
Title: The Effect of Gamification on Disease Self-Management and Glycemic Control in Patients With Type 2 Diabetes
Brief Title: The Effect of Gamification on Patients With Type 2 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sakarya University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: SakaryaU.
Record Dates: First submitted 2022-12-22; First posted 2023-02-13 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Gamification; Type 2 Diabetes; Self-management; Digital Health; Mobile Application
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Application of data collection forms for the initial evaluation. Teaching the use of mobile games, monitoring the use of mobile games in the experimental group by the researcher for six weeks, and applying data collection forms to the patients in the sixth week.
  Interventions: Other: Gamification and education with mobile game application
- Control Group (No Intervention): Application of data collection forms for the initial evaluation. Application of data collection forms to the patients in the sixth week. No intervention will be made to the patients in the control group other than the routine education given in the diabetes outpatient clinic.

INTERVENTIONS:
Other: Gamification and education with mobile game application — This study aimed to provide self-care management by playing mobile games to patients with type 2 diabetes.
  Arms: Intervention Group

SUMMARY:
Diabetes is a broad-spectrum metabolic disorder that causes a defect in the organism's carbohydrate, fat, and protein metabolism processes due to insulin deficiency or impaired insulin effect. Diabetes requires continuous medical care and causes chronic, severe mortality and morbidity. More than 90% of all people with diabetes worldwide suffer from Type 2 DM. Diabetes self-management includes self-monitoring of blood glucose levels, knowing and managing the symptoms of hypoglycemia and hyperglycemia, adherence to diet, physical exercise, and diabetic foot care. Considering the high prevalent and undesirable consequences of diabetes in the world, it is necessary to benefit from new educational technologies and tools. One of these technologies is gamification, which increases the quality of education as an effective educational tool, creates motivation and enthusiasm, and develops a sense of competition in the target audience. This study plans to develop a game that will include virtual coaching to increase the self-management and glycemic control of patients with type 2 diabetes.

DETAILED DESCRIPTION:
The research will be carried out in two stages. In Stage 1, the game will be developed; The developed game's effectiveness will be evaluated in the 2nd stage by testing it. The game's content will include healthy nutrition, exercise, foot care, insulin use, and hypoglycemia management. When the games are completed, the virtual coach will step in, and the participants will be given motivational feedback. The game developed will be evaluated by the patients in the second stage with a two-week pilot period. It will be updated according to the feedback received. The final version of the game will be passed forward to the implementation phase. Individuals who are willing to participate in the study coming to Prof. Dr. Cemil Tascioglu City Hospital Diabetes Polyclinic will be randomly assigned to the intervention and control groups. A total of 88 patients (44 controls - 44 experiments) are planned to be recruited. In the first interview with the individuals in the intervention group, Within the scope of the pretest, the "Personal Information Form," "Anthropometric Measurement Form," "Metabolic Control Variables Form," and "Diabetes Self-Management Scale" will be used for evaluation. Outpatient appointment dates of the sixth week of the intervention program, "Anthropometric Measurement Form," "Metabolic Control Variables Form," and "Diabetes Self-Management Scale" forms will be used with patients for the final evaluation within the scope of the posttest.

In the first meeting with the individuals in the control group, explanations about the research will be made. After their written consent is obtained at the first interview and within the scope of the pretest, the "Personal Information Form," "Anthropometric Measurement Form," "Metabolic Control Variables Form," and "Diabetes Self-Management Scale" will be used for evaluation. At the end of the sixth week of the study, when they come in for their outpatient clinic appointments, as a part of the posttest, "Anthropometric Measurement Form," "Metabolic Control Variables Form," and "Diabetes Self-Management Scale" forms will be used for the final evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Two years or more with a diagnosis of Type 2 DM
* Patients using Insulin or Insulin and Oral Antidiabetic
* No sensory loss, such as vision and hearing loss,
* Having internet access and being able to use it,
* Ability to use a mobile phone with an Android or IOS (iPhone OS) operating system
* Patients who agreed to participate in the study

Exclusion Criteria:

* Patients diagnosed with Type 1 DM and Gestational DM.
* Visual and auditory loss,
* Individuals without internet access
* Unable to communicate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2023-02-25 (Estimated); Primary Completion 2023-09-17 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
self-management scale | Change between the first day and the sixth week of the study
  Determining whether or not the disease self-management scale scores in patients with Type 2 DM using the developed mobile game application increased at the end of the 6 weeks period. A minimum of 0 and a maximum of 10 points are obtained on the scale. If an item is skipped, it is evaluated as -3 points. Diabetes self-management increases as the score get closer to 10.

SECONDARY OUTCOMES:
glycemic control (HbA1c) | Change between day one and week 6 of the study
  The effect that the mobile game application developed imposes on glycemic control in patients with Type 2 DM at six weeks compared to baseline.
  The effect of the patient's HbA1c tests on the 6th week compared to the baseline.
  Blood test (HbA1c) will be performed during the outpatient follow-up at the first and sixth weeks.
anthropometric measurements (Body Mass Index) | The change between the first day and the sixth week of the study
  The effects on anthropometric measurements in patients with Type 2 DM using the mobile game application developed compared to baseline at week 6.
  The effect on the patient's Body Mass Index compared to baseline at week 6. The researcher will measure it.
  Body Mass Index is calculated by dividing the person's weight in kilograms by the square of the person's height in meters (kg/m²).

CONTACTS AND LOCATIONS:
Locations (1):
- Pelin ILHAN, Istanbul, Sisli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No